CLINICAL TRIAL: NCT04080544
Title: Cause or Effect: Untangling the Relationship With Amyloid and Tau Deposits to Cognitive Decline and Alzheimer's Disease in the Dallas Lifespan Brain Study
Brief Title: Cognitive Decline and Alzheimer's Disease in the Dallas Lifespan Brain Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Neil M Rofsky, MD, MHA (Other)
Responsible Party: Sponsor-Investigator, Neil M Rofsky, MD, MHA, Professor and Chair, Department of Radiology, University of Texas Southwestern Medical Center
Organization: University of Texas Southwestern Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 092015-003
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-08

CONDITIONS: Alzheimer Disease; Cognitive Decline
Keywords: Positron Emission Tomography
MeSH Terms: conditions — Alzheimer Disease; Cognitive Dysfunction | interventions — 7-(6-fluoropyridin-3-yl)-5H-pyrido(4,3-b)indole; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Follow up DLBS participants (Experimental): Eight to ten year follow-up DLBS participants who were cognitively normal at the time of enrollment from 2008 to 2014.
  Interventions: Drug: [18F]AV-1451; Procedure: Positron Emission Tomography

INTERVENTIONS:
Drug: [18F]AV-1451 — The subject will receive up to a target dose of 370 megabecquerel (MBq) as a single IV bolus of [18F]AV-1451.
  Other Names: Flortaucipir F18
Procedure: Positron Emission Tomography — Approximately 80 minutes after injection subjects will be placed in the UTSW PET/CT scanner for a 20-minute brain scan.
  Other Names: PET

SUMMARY:
The investigators will conduct tau positron emission tomography (PET) scans on 125 adults using the radiopharmaceutical Flortaucipir F18 ([18F]AV-1451). This will allow the investigators to determine tau deposition across adults of different ages and assess the relationship of current tau burden to cognitive function and amyloid deposition collected over the previous 10-year interval.

DETAILED DESCRIPTION:
Alzheimer's disease (AD) is a highly prevalent disorder of dementia in older adults. AD neuropathology is marked by the presence of amyloid plaques and tau neurofibrillary tangles. Autopsy studies, as well as magnetic resonance imaging (MRI) studies in living persons, have established that the neurodegenerative changes in AD begin in medial temporal lobe structures and later progress to adjacent temporal, parietal and frontal neocortical regions. Magnetic resonance image studies of AD consistently reveal volumetric loss in the hippocampus using both cross-sectional and longitudinal approaches. The primary symptom of early-stage AD is memory impairment possibly accompanied by deficits in attentional control. Normal aging, however, is also marked by cognitive decline, as well as structural brain changes. Autopsy data had shown in the past that about 30% of older adults with no obvious cognitive impairment show some degree of the neuropathology typically associated with dementia at autopsy.

Importantly, the recent ability to image beta-amyloid and tau deposits in vivo using positron emission tomography (PET) scanning has revolutionized our understanding of early stages of AD. Evidence suggests that amyloid deposits may be detected 10 - 15 years before memory symptoms appear. These findings are leading to the ability to diagnose AD years before symptoms begin. Much less is known about the impact and developmental course of tau deposition as compared to beta-amyloid because the ligand to image tau was only recently invented. There is increasing evidence that tau is particularly toxic to the brain and is a later precursor of AD than amyloid deposits. Additional research on beta-amyloid and tau deposition in aging is crucial, as much work suggests that treatment of AD may be most effective when implemented early in the time course of the disease. Understanding the impact of tau deposits and its interactions with amyloid deposition allows the investigators to see the development of early markers of AD, which are important in understanding the trajectory of the disease. An important approach to understand the amyloid/tau puzzle and its relationship to AD is a large-scale longitudinal study of normal aging that integrates extensive neuroimaging and cognitive assessments along with tau imaging. A key aspect in understanding pathological aging is the need to be able to clearly differentiate normal aging from early pathology. The present Tau imaging study described here is an important component of the Dallas Lifetime Brain Study (DLBS).

The Dallas Lifespan Brain Study (DLBS) began in 2008 and was designed to utilize the new in vivo imaging techniques to address uncertainty regarding how AD pathology relates to the developmental process of aging and cognition, fueled in part by the partial overlap of pathological markers and decline in mnemonic function observed in a substantial proportion of 'normal' aged individuals. A total of 296 participants were recruited for Wave 1 from 2008 to 2014 to the DLBS and they received cognitive testing, structural and functional MRI, as well as a scan for beta amyloid using the radioligand AV-45 Florbetapir F 18 (also known as "[18F]AV-45"). A total of 183 returning participants were tested four years later in Wave 2, and they received the same battery as in Wave 1. In addition, 60 of these were also scanned with Flortaucipir F 18 (also known as "[18F]AV-1451"). [18F]AV-1451 is a newly-developed Phase II ligand that measures tau deposit in the human brain and this drug was provided to the DLBS by Avid Radiopharmaceuticals.

The objective of the current study is to test 125 DLBS participants with [18F]AV-1451 (Flortaucipir F 18) at the University of Texas Southwestern Medical Center (UTSW). The inclusion of tau imaging in Wave 3 will allow the investigators to relate tau deposition in the brain to the 10-year history of amyloid deposition and cognitive decline in the DLBS participants and understand the independent and joint contributions of tau to cognitive decline and early AD at different ages.

ELIGIBILITY:
Inclusion Criteria:

* Participated in Wave 1 or 2 of the DLBS study.
* Subjects must indicate that they are not currently pregnant if they are women of child-bearing potential. Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 90 days following completion of therapy. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A female of child-bearing potential is any woman (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria: 1) Has not undergone a hysterectomy or bilateral oophorectomy; or 2) Has not been naturally post-menopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
* Volumetric Brain MRI Image (T-1 Weighted MPRage) collected as part of DLBS Wave 1, 2, or 3 protocol.
* Completed at least 9 years of formal education, or the equivalent of freshman year of high school.
* Fluent English speakers.
* Tolerate laying 20 minutes on a flat table for the PET scan.
* Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Mini-Mental State Examination (MMSE) score lower than 22; all DLBS participants at the time of initial Wave 1 enrollment between 2008 - 2014 had an MMSE score of 26 or above, indicating normal cognitive function. However, in the time interval between Wave 1 and Wave 3, it is possible that mental capacity may have deteriorated. The investigators will exclude all participants in Wave 3 testing who have an MMSE lower than 22.
* Taking some types of sedatives, benzodiazepines, or anti-psychotics.
* Currently undergoing chemotherapy or radiation for cancer.
* New history of substance abuse.
* Has a history of drug or alcohol dependence within the last year, or prior prolonged history of dependence.
* Recreational drug use in past six months.
* Central nervous systems disease or brain injury that would preclude participation in the study.
* Psychiatric or neurological disorder that would preclude participation in this study.
* Has clinically significant hepatic, renal, pulmonary, metabolic or endocrine disturbances which pose safety risk.
* Has a current clinically significant cardiovascular disease that poses a safety risk.
* Has a current clinically significant infectious disease or a medical comorbidity which poses a safety risk.
* Has either: 1) Screening electrocardiogram (ECG) with corrected QT Interval (QTc) > 450 millisecond (msec) if male, or QTc > 470 msec if female; or 2) A history of additional risk factors for Torsades de Pointes (TdP) (e.g., hypokalemia, family history of Long QT syndrome) or are taking drugs that are known to cause QT prolongation (a list of prohibited and discouraged medications is provided by the Sponsor); Patients with a prolonged QTc interval in the setting of intraventricular conduction block (examples right bundle branch block or left bundle branch block), may be enrolled with sponsor approval.
* Has received or will receive investigational medication within the 30 days of PET/CT scan.
* Has received or will receive a radiopharmaceutical for imaging or therapy within 24 hours of PET/CT scan.
* Is a participant who, in the opinion of the investigator(s), is otherwise unsuitable for a study of this type.

Ages: 38 Years to 96 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-01-15 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Denise Park, PhD, Principal Investigator — The University of Texas at Dallas
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Balota D.A., Faust M.E. (2001). Attention in dementia of the Alzheimer's type. In: Boller F, Cappa S, editors. Handbook of Neuropsychology. 2nd Ed. NY: Elsevier Science; pp. 51-80.
- [Background] Bennett DA, Schneider JA, Tang Y, Arnold SE, Wilson RS. The effect of social networks on the relation between Alzheimer's disease pathology and level of cognitive function in old people: a longitudinal cohort study. Lancet Neurol. 2006 May;5(5):406-12. doi: 10.1016/S1474-4422(06)70417-3. PMID 16632311
- [Background] Braak H, Braak E. Neuropathological stageing of Alzheimer-related changes. Acta Neuropathol. 1991;82(4):239-59. doi: 10.1007/BF00308809. PMID 1759558
- [Background] Convit A, de Leon MJ, Golomb J, George AE, Tarshish CY, Bobinski M, Tsui W, De Santi S, Wegiel J, Wisniewski H. Hippocampal atrophy in early Alzheimer's disease: anatomic specificity and validation. Psychiatr Q. 1993 Winter;64(4):371-87. doi: 10.1007/BF01064929. PMID 8234547
- [Background] Holm S: A Simple Sequentially Rejective Bonferroni Test. Scandinavian Journal of Statistics. 1979, 65 -670.
- [Background] Kemper S, Anagnopoulos C, Lyons K, Heberlein W. Speech accommodations to dementia. J Gerontol. 1994 Sep;49(5):P223-9. doi: 10.1093/geronj/49.5.p223. PMID 8056947
- [Background] Khachaturian ZS. Diagnosis of Alzheimer's disease. Arch Neurol. 1985 Nov;42(11):1097-105. doi: 10.1001/archneur.1985.04060100083029. No abstract available. PMID 2864910
- [Background] Killiany RJ, Moss MB, Albert MS, Sandor T, Tieman J, Jolesz F. Temporal lobe regions on magnetic resonance imaging identify patients with early Alzheimer's disease. Arch Neurol. 1993 Sep;50(9):949-54. doi: 10.1001/archneur.1993.00540090052010. PMID 8363449
- [Background] Jack, C., Knopman, D., Jagust, W., Petersen, R., Weiner, M., Aisen, P., … Trojanowski, J. (2013). Update on hypothetical model of Alzheimer's disease biomarkers. Alzheimer's & Dementia, 9(4), 521-522.
- [Background] Jack CR Jr, Petersen RC, Xu YC, Waring SC, O'Brien PC, Tangalos EG, Smith GE, Ivnik RJ, Kokmen E. Medial temporal atrophy on MRI in normal aging and very mild Alzheimer's disease. Neurology. 1997 Sep;49(3):786-94. doi: 10.1212/wnl.49.3.786. PMID 9305341
- [Background] Mohs RC, Ashman TA, Jantzen K, Albert M, Brandt J, Gordon B, Rasmusson X, Grossman M, Jacobs D, Stern Y. A study of the efficacy of a comprehensive memory enhancement program in healthy elderly persons. Psychiatry Res. 1998 Feb 27;77(3):183-95. doi: 10.1016/s0165-1781(98)00003-1. PMID 9707301
- [Background] Park DC, Reuter-Lorenz P. The adaptive brain: aging and neurocognitive scaffolding. Annu Rev Psychol. 2009;60:173-96. doi: 10.1146/annurev.psych.59.103006.093656. PMID 19035823
- [Background] Price JL, Ko AI, Wade MJ, Tsou SK, McKeel DW, Morris JC. Neuron number in the entorhinal cortex and CA1 in preclinical Alzheimer disease. Arch Neurol. 2001 Sep;58(9):1395-402. doi: 10.1001/archneur.58.9.1395. PMID 11559310
- [Background] Reuter-Lorenz PA, Park DC. How does it STAC up? Revisiting the scaffolding theory of aging and cognition. Neuropsychol Rev. 2014 Sep;24(3):355-70. doi: 10.1007/s11065-014-9270-9. Epub 2014 Aug 21. PMID 25143069
- [Background] Sperling RA, Aisen PS, Beckett LA, Bennett DA, Craft S, Fagan AM, Iwatsubo T, Jack CR Jr, Kaye J, Montine TJ, Park DC, Reiman EM, Rowe CC, Siemers E, Stern Y, Yaffe K, Carrillo MC, Thies B, Morrison-Bogorad M, Wagster MV, Phelps CH. Toward defining the preclinical stages of Alzheimer's disease: recommendations from the National Institute on Aging-Alzheimer's Association workgroups on diagnostic guidelines for Alzheimer's disease. Alzheimers Dement. 2011 May;7(3):280-92. doi: 10.1016/j.jalz.2011.03.003. Epub 2011 Apr 21. PMID 21514248
- [Background] Storandt M, Grant EA, Miller JP, Morris JC. Rates of progression in mild cognitive impairment and early Alzheimer's disease. Neurology. 2002 Oct 8;59(7):1034-41. doi: 10.1212/wnl.59.7.1034. PMID 12370458
- [Background] Trojanowski JQ, Clark CM, Schmidt ML, Arnold SE, Lee VM. Strategies for improving the postmortem neuropathological diagnosis of Alzheimer's disease. Neurobiol Aging. 1997 Jul-Aug;18(4 Suppl):S75-9. doi: 10.1016/s0197-4580(97)00075-4. PMID 9330990
- [Background] Whalley LJ. Brain ageing and dementia: what makes the difference? Br J Psychiatry. 2002 Nov;181:369-71. doi: 10.1192/bjp.181.5.369. No abstract available. PMID 12411259

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Scans were acquired from participants previously enrolled in Wave 1 or 2 of the Dallas Lifespan Brain Study (DLBS)
Groups:
- Follow up DLBS Participants: Eight to ten year follow-up DLBS participants who were cognitively normal at the time of enrollment from 2008 to 2014.
  [18F]AV-1451: The subject will receive up to a target dose of 370 megabecquerel (MBq) as a single IV bolus of [18F]AV-1451.
  Positron Emission Tomography: Approximately 80 minutes after injection subjects will be placed in the University of Texas Southwestern Medical Center (UTSW) Positron Emission Tomography/Computed Tomography (PET/CT) scanner for a 20-minute brain scan.
Period: Overall Study
Arm/Group | Follow up DLBS Participants
Started | 125
Completed | 125
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 49
  >=65 years | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.70 (14.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77
  Male | 48
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6
  Not Hispanic or Latino | 119
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 112
  More than one race | 5
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 125
Education, Continuous [Mean (Standard Deviation); unit: years] | 16.09 (2.10)
Mini-Mental State Examination [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental State Examination (MMSE) is a simple pen-and-paper test of cognitive function. The total score is reported (range: 0-30 points) and higher scores on the MMSE reflect better cognitive function.
  units on a scale | 28.36 (1.50)

OUTCOME MEASURES:

1. Primary Outcome: Standardized Uptake Value Ratios (SUVrs) Calculated From [18F]AV-1451 PET Scans
Description: Tau accumulation in the temporal lobe will be measured as the standardized uptake value ratio (SUVR) computed from each participant's [18F]AV-1451 PET scans averaged across six bilateral regions of interest (ROls) by normalizing regional counts to the whole cerebellum. The 6 ROls are: inferior temporal gyrus, middle temporal gyrus, superior temporal gyrus, entorhinal cortex, parahippocampal gyrus, and fusiform gyrus. Each participant's PET scan and the six bilateral ROIs will be coregistered to their T1-weighted MRI (MP-RAGE). Finally, the mean observed tracer count from each region will be extracted and normalized using whole cerebellum as the reference. Observed tau SUVR scores in humans range from 0.5 to 2.5, with higher scores being indicative of greater tau accumulation. Unless otherwise specified, all subsequent analyses will use this temporal tau SUVR and will involve examination of cross-sectional relationships between tau SUVR and key outcome measures at Wave 3 of the DLBS.
Time Frame: An average of 3-months post-PET study visit
Population: Participants with available data were analyzed. This sample excludes one participant whose scanner data were unusable due to technical issues during acquisition.
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 124
standardized uptake value ratio | 1.09 (0.10)

2. Secondary Outcome: Relationship of Tau Burden to Episodic Memory Function
Description: Episodic memory is a construct that measures how well individuals can store, maintain, and retrieve detailed information in long-term memory. Episodic memory will be a composite score using the Hopkins Verbal Learning test with 3 subcomponents (immediate recall: range 0-12, delayed recall: range 0-12, and recognition: range 0-24) and the immediate recall of the CANTAB Verbal Recognition Memory task (range 0-12). Scores from the tasks will be converted to Z-scores and averaged to form an episodic memory composite, and then this final value with be converted to a Z-score. A higher composite Z-score indicates better episodic memory, a Z-score of 0 represents the population mean, and all Z-scores have a standard deviation of 1. Values in this table represent this Episodic Memory Z-score.
Time Frame: 1-year post study completion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 124
Z-score | 0 (1)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to episodic memory; Test type: Other — Null-hypothesis significance testing; p = .081, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = -1.42, 95% CI 2-sided [-3.03 to 0.18], Standard Error of Mean 0.81
Statistical Analysis 2: Comparison: Follow up DLBS Participants; Regression testing the interaction of temporal tau SUVR and amyloid SUVR in prediction of episodic memory; Test type: Other — Null-hypothesis significance test; p = .604, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = -0.07, 95% CI 2-sided [-0.32 to 0.19], Standard Error of Mean 0.13

3. Secondary Outcome: Relationship of Amyloid Accumulation to Tau Burden
Description: Amyloid accumulation throughout the Dallas Lifespan Brain Study (6-9.8 years) will be measured with Florbetapir F18 and calculated as an Amyloid Standard Uptake Value ratio (SUVR) by normalizing regional counts to the whole cerebellum. Amyloid SUVR scores will be averaged across eight cortical regions spanning most of the cortex: dorsal lateral prefrontal cortex, orbitofrontal cortex, lateral parietal cortex, posterior cingulate cortex, anterior cingulate cortex, precuneus, lateral temporal cortex, and lateral occipital lobe. Amyloid SUVR scores observed in this study have ranged from 0.88 to 1.74, with higher scores being indicative of greater amyloid accumulation. Finally, annualized change scores for these amyloid SUVRs across the full study duration (6-9.8 years) will be calculated to determine the extent that the rate of amyloid accumulation relates to tau burden at the end of the study.
Time Frame: 1-year post study completion
Population: Participants with available data were analyzed.
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 59
standardized uptake value ratio | 0.0035 (0.0122)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship between amyloid accumulation (annualized change score for amyloid SUVR) to temporal tau SUVR; Test type: Other — Null-hypothesis significance test; p = .033, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for baseline age, sex, and years of education; Slope = 1.77, 95% CI 2-sided [0.15 to 3.39], Standard Error of Mean 0.81

4. Secondary Outcome: Relationship of Tau Burden to Speed of Processing
Description: Speed of processing is a construct that measures how rapidly individuals can process information. To assess speed of processing, a composite score will be created using the Digit Comparison task and the Wechsler Adult Intelligence Scale (WAIS) Digit Symbol task. Observed DLBS raw scores range from 27 to 116 for Digit Comparison task and 20 to 90 for Digit Symbol task. Participants' raw scores are converted to Z-scores and averaged to form a speed of processing composite, and then this final value with be converted to a Z-score. A higher composite Z-score indicates better speed of processing, a Z-score of 0 represents the population mean, and all Z-scores have a standard deviation of 1. Values in this table represent this Speed of Processing Z-score.
Time Frame: 1-year post study completion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 124
Z-score | 0 (1)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to speed of processing; Test type: Other — Null-hypothesis significance testing; p = .699, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = .272, 95% CI 2-sided [-1.12 to 1.66], Standard Error of Mean .70
Statistical Analysis 2: Comparison: Follow up DLBS Participants; Regression testing the interaction of temporal tau SUVR and amyloid SUVR in the prediction of speed of processing; Test type: Other — Null-hypothesis significance test; p = .154, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.16, 95% CI 2-sided [-0.06 to 0.38], Standard Error of Mean 0.11

5. Secondary Outcome: Relationship of Tau Burden to Reasoning
Description: The construct of reasoning measures an individual's ability to recognize novel patterns and the conceptual relationship among objects and effectively apply these patterns to solve similar problems. To assess reasoning, a composite score will be created using the Raven's Progressive Matrices task and Educational Testing Service (ETS) Letters Sets task. Observed DLBS raw scores range from 9 to 30 for Raven's Progressive Matrices task and from 0.5 to 30 for ETS Letters Sets task. Raven's Progress Matrices and ETS Letter Sets will be converted to Z-scores and averaged to form a reasoning composite, and then this final value with be converted to a Z-score. A higher composite Z-score indicates higher reasoning ability, a Z-score of 0 represents the population mean, and all Z-scores have a standard deviation of 1. Values in this table represent this Reasoning Z-score.
Time Frame: 1-year post study completion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-scores
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 124
Z-scores | 0 (1)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to reasoning function; Test type: Other — Null-hypothesis significance testing; p = .137, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = -1.11, 95% CI 2-sided [-2.58 to 0.36], Standard Error of Mean 0.74
Statistical Analysis 2: Comparison: Follow up DLBS Participants; Regression testing the interaction of temporal tau SUVR and amyloid SUVR in prediction of reasoning; Test type: Other — Null-hypothesis significance test; p = .428, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.11, 95% CI 2-sided [-0.16 to 0.37], Standard Error of Mean 0.13

6. Secondary Outcome: Relationship of Tau Burden to Working Memory
Description: Working memory is a construct that measures the ability of individuals to simultaneously manipulate and store information. To assess working memory, a composite score will be created using the CANTAB Spatial Working Memory task (reverse scored) and the Wechsler Adult Intelligence Scale (WAIS-III) Letter Number Sequencing task. Observed DLBS raw scores range from 0 to 86 total errors for the CANTAB Spatial Working Memory task and 2 to 20 for the WAIS-III Letter Number Sequencing task. Participants' raw scores are converted to Z-scores and averaged to form a working memory composite, and then this final value with be converted to a Z-score. A higher working memory composite Z-score indicates better working memory, a Z-score of 0 represents the population mean, and all Z-scores have a standard deviation of 1. Values in this table represent this Working Memory Z-score.
Time Frame: 1-year post study completion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 124
Z-score | 0 (1)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to working memory; Test type: Other — Null-hypothesis significance test; p = .376, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = -0.70, 95% CI 2-sided [-2.25 to 0.86], Standard Error of Mean 0.78
Statistical Analysis 2: Comparison: Follow up DLBS Participants; Regression testing the interaction of temporal tau SUVR and amyloid SUVR in prediction of working memory; Test type: Other — Null-hypothesis significance test; p = .039, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.27, 95% CI 2-sided [0.01 to 0.53], Standard Error of Mean 0.13
Statistical Analysis 3: Comparison: Follow up DLBS Participants; Post hoc simple slopes test of the amyloid x tau interaction (Statistical Analysis #2) at 1SD below the mean for amyloid; Test type: Other — Null-hypothesis significance test; p = .091, sim_slopes (R interactions package) — A priori threshold was two-sided 0.017 after Bonferroni correction for multiple comparisons (3 post hoc tests); Slope = -0.47, Standard Error of Mean 0.27
Statistical Analysis 4: Comparison: Follow up DLBS Participants; Post hoc simple slopes test of the amyloid x tau interaction (Statistical Analysis #2) at the mean for amyloid SUVR; Test type: Other — Null-hypothesis significance test; p = .296, sim_slopes (R interactions package) — A priori threshold was two-sided 0.017 after Bonferroni correction for multiple comparisons (3 post hoc tests); Slope = -0.20, Standard Error of Mean 0.19
Statistical Analysis 5: Comparison: Follow up DLBS Participants; Post hoc simple slopes test of the amyloid x tau interaction (Statistical Analysis #2) at 1SD above the mean for amyloid SUVR; Test type: Other — Null-hypothesis significance test; p = .695, sim_slopes (R interactions package) — A priori threshold was two-sided 0.017 after Bonferroni correction for multiple comparisons (3 post hoc tests); Slope = 0.07, Standard Error of Mean 0.17

7. Secondary Outcome: Relationship of Tau Burden to Participants' Age
Description: Linear regressions between the AV-1451 SUVR in each of the temporal regions of interest with participant age will be calculated, and in additional analyses, non-linear effects of age will be examined via quadratic and growth modeling. Observed AV-1451 SUVR scores in humans have ranged from 0.5 to 2.5, with higher scores being indicative of greater tau accumulation. The investigators predict that tau accumulation will accelerate in old age, thus supporting a non-linear rate of deposition.
Time Frame: 1-year post study completion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: standardized uptake value ratio
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 124
standardized uptake value ratio
  inferior temporal SUVR | 1.14 (0.13)
  middle temporal SUVR | 1.11 (0.13)
  superior temporal SUVR | 1.04 (0.07)
  entorhinal SUVR | 1.09 (0.14)
  parahippocampal SUVR | 1.05 (0.10)
  fusiform SUVR | 1.13 (0.08)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(linear) to inferior temporal SUVR; Test type: Other — Null-hypothesis significance test; p = .012, Regression, Linear — A prior threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.002, 95% CI 2-sided [0.0004 to 0.004], Standard Error of Mean 0.001
Statistical Analysis 2: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(quadratic) to inferior temporal SUVR; Test type: Other — Null-hypothesis significance test; p = .905, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = -0.000005, 95% CI 2-sided [-0.000009 to 0.00008], Standard Error of Mean 0.00004
Statistical Analysis 3: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(growth model) to inferior temporal SUVR. Growth modeling was performed using SPSS curve estimation; Test type: Other — Null-hypothesis significance test; p = .006, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.002, Standard Error of Mean 0.001
Statistical Analysis 4: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(linear) to middle temporal gyrus SUVR; Test type: Other — Null-hypothesis significance test; p = .018, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.002, 95% CI 2-sided [0.0003 to 0.003], Standard Error of Mean 0.001
Statistical Analysis 5: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(quadratic) to middle temporal SUVR; Test type: Other — Null-hypothesis significance test; p = .579, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustment for multiple comparisons; Slope = -0.00002, 95% CI 2-sided [-0.0001 to 0.00006], Standard Error of Mean 0.00004
Statistical Analysis 6: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(growth model) to middle temporal SUVR. Growth modeling was performed using SPSS curve estimation; Test type: Other — Null-hypothesis significance test; p = .008, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.002, Standard Error of Mean 0.001
Statistical Analysis 7: Comparison: Follow up DLBS Participants; Regression testing the relationship of age to superior temporal SUVR; Test type: Other — Null-hypothesis significance test; p = .897, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.00006, 95% CI 2-sided [-0.001 to 0.001], Standard Error of Mean 0.0004
Statistical Analysis 8: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(quadratic) to superior temporal SUVR; Test type: Other — Null-hypothesis significance test; p = .539, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = -0.00002, 95% CI 2-sided [-0.00007 to 0.00003], Standard Error of Mean 0.00003
Statistical Analysis 9: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(growth model) to superior temporal SUVR. Growth modeling was performed using SPSS curve estimation; Test type: Other — Null-hypothesis significance test; p = .973, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = -0.00001, Standard Error of Mean 0.0004
Statistical Analysis 10: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(linear) to entorhinal SUVR; Test type: Other — Null-hypothesis significance test; p = .200, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.001, 95% CI 2-sided [-0.001 to 0.003], Standard Error of Mean 0.001
Statistical Analysis 11: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(quadratic) to entorhinal SUVR; Test type: Other — Null-hypothesis significance test; p = .346, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.00005, 95% CI 2-sided [-0.00005 to 0.0001], Standard Error of Mean 0.00005
Statistical Analysis 12: Comparison: Follow up DLBS Participants; Regression testing relationship of age(growth model) to entorhinal SUVR. Growth modeling was performed using SPSS curve estimation; Test type: Other — Null-hypothesis significance test; p = .283, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.001, Standard Error of Mean 0.001
Statistical Analysis 13: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(linear) to parahippocampal SUVR; Test type: Other — Null-hypothesis significance test; p = .011, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.002, 95% CI 2-sided [0.0004 to 0.003], Standard Error of Mean 0.001
Statistical Analysis 14: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(quadratic) to parahippocampal SUVR; Test type: Other — Null-hypothesis significance test; p = .536, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.00002, 95% CI 2-sided [-0.00004 to 0.00009], Standard Error of Mean 0.00003
Statistical Analysis 15: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(growth model) to parahippocampal SUVR. Growth modeling was performed using SPSS curve estimation; Test type: Other — Null-hypothesis significance test; p = .013, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.001, Standard Error of Mean 0.001
Statistical Analysis 16: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(linear) to fusiform SUVR; Test type: Other — Null-hypothesis significance test; p < .001, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.002, 95% CI 2-sided [0.001 to 0.003], Standard Error of Mean 0.0005
Statistical Analysis 17: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(quadratic) to fusiform SUVR; Test type: Other — Null-hypothesis significance test; p = .692, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.00001, 95% CI 2-sided [-0.00004 to 0.00006], Standard Error of Mean 0.00003
Statistical Analysis 18: Comparison: Follow up DLBS Participants; Regression testing the relationship of age(growth model) to fusiform SUVR. Growth modeling was performed using SPSS curve estimation; Test type: Other — Null-hypothesis significance test; p < .001, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; No adjustments were made; Slope = 0.001, Standard Error of Mean 0.0004

8. Secondary Outcome: Relationship of Tau Burden to Cortical Thickness
Description: Regional cortical thickness will be estimated from previously acquired T1-weighted structural magnetic resonance imaging (MRl) scans using FreeSurfer (ver. 5.3), with surface parcellation manually edited when necessary by our team of experts. The regions selected for analyses of cortical thickness were the ROIs used to estimate temporal tau SUVR: inferior temporal gyrus, middle temporal gyrus, superior temporal gyrus, entorhinal cortex, parahippocampal gyrus, and fusiform gyrus. Observed cortical thickness in these regions range from 1.38 to 3.83 mm with higher scores indicating greater thickness.
Time Frame: 1-year post study completion
Population: Participants with available data were analyzed. This sample excludes one participant whose scanner data were unusable due to technical issues during acquisition and three participants did not have a recent MRI.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 121
mm
  inferior temporal thickness | 2.53 (0.22)
  middle temporal thickness | 2.68 (0.20)
  superior temporal thickness | 2.51 (0.25)
  parahippocampal thickness | 2.44 (0.26)
  entorhinal thickness | 2.85 (0.47)
  fusiform thickness | 2.46 (0.21)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to inferior temporal gyrus cortical thickness; Test type: Other — Null-hypothesis significance testing; p = .331, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.18, 95% CI 2-sided [-0.18 to 0.53], Standard Error of Mean 0.18
Statistical Analysis 2: Comparison: Follow up DLBS Participants; Regression testing the relationship between temporal tau SUVR to middle temporal gyrus cortical thickness; Test type: Other — Null-hypothesis significance testing; p = .636, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.07, 95% CI 2-sided [-0.24 to 0.39], Standard Error of Mean 0.16
Statistical Analysis 3: Comparison: Follow up DLBS Participants; Regression testing the relationship between temporal tau SUVR to superior temporal gyrus cortical thickness; Test type: Other — Null-hypothesis significance testing; p = .024, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.38, 95% CI 2-sided [0.05 to 0.70], Standard Error of Mean 0.16
Statistical Analysis 4: Comparison: Follow up DLBS Participants; Regression testing the relationship between temporal tau SUVR to parahippocampal gyrus cortical thickness; Test type: Other — Null-hypothesis significance testing; p = .235, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = -0.27, 95% CI 2-sided [-0.73 to 0.18], Standard Error of Mean 0.23
Statistical Analysis 5: Comparison: Follow up DLBS Participants; Regression testing the relationship between temporal tau SUVR to entorhinal gyrus cortical thickness; Test type: Other — Null-hypothesis significance testing; p = .639, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.19, 95% CI 2-sided [-0.63 to 1.01], Standard Error of Mean 0.41
Statistical Analysis 6: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to fusiform gyrus cortical thickness; Test type: Other — Null-hypothesis significance test; p = .252, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.19, 95% CI 2-sided [-0.13 to 0.50], Standard Error of Mean 0.16

9. Secondary Outcome: Relationship of Tau Burden to Hippocampal Volume
Description: Hippocampal volume will be estimated from previously acquired T1-weighted structural magnetic resonance imaging (MRl) scans using FreeSurfer (ver. 5.3), with surface parcellation manually edited when necessary by our team of experts. This region was selected for analysis as it was one of the ROIs used to estimate temporal tau SUVR. Observed DLBS hippocampal volume ranged from 1843 to 5342 mm^3 with higher scores indicating greater volume.
Time Frame: 1-year post study completion
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 121
mm^3 | 3864.98 (626.45)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to hippocampal volume; Test type: Other — Null-hypothesis significance test; p = .619, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = -233.74, 95% CI 2-sided [-1163.28 to 695.79], Standard Error of Mean 469.31

10. Secondary Outcome: Relationship of Tau Burden to White Matter Integrity
Description: White matter integrity will be assessed using the estimated volume of white matter hypointensities from previously acquired T1-weighted structural magnetic resonance imaging (MRl) scans using FreeSurfer (ver. 5.3). Observed DLBS white matter hypointensities range from 796 to 35,037 mm^3 with higher scores indicating greater volume of hypointensities and reflecting worse white matter integrity.
Time Frame: 1-year post study completion
Population: Participants with available data were analyzed. This sample excludes one participant whose scanner data were unusable due to technical issues during acquisition and three participants who did not have a recent MRI.
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 121
mm^3 | 3864.48 (4539.80)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to volume of white matter hypointensities; Test type: Other — Null-hypothesis significance test; p = .017, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 9260.01, 95% CI 2-sided [1660.52 to 16859.51], Standard Error of Mean 3836.92

11. Secondary Outcome: Relationship of Tau Burden to Functional Magnetic Resonance Imaging (MRI)
Description: For functional measures, blood oxygenation level dependent signal from contrasts of interest using selected ROls will be created. For the semantic judgment task (easy judgments - fixation), the investigators will focus on ROIs associated with processing meaning, including inferior frontal gyrus, precuneus, and middle temporal gyrus. Observed BOLD activation values (betas) ranged from -1.00 to 1.30 with higher values indicating greater activation.
Time Frame: 1-year post study completion
Population: Participants with available tau and fMRI data were analyzed.
Measure: Mean (Standard Deviation); unit: fMRI activation beta
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 98
fMRI activation beta
  Inferior frontal gyrus | 0.27 (0.31)
  Middle temporal gyrus | 0.07 (0.26)
  Precuneus | -0.23 (0.36)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to activation of inferior frontal gyrus (beta) on the semantic judgment fMRI task; Test type: Other — Null-hypothesis significance test; p = .411, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.29, 95% CI 2-sided [-0.41 to 0.99], Standard Error of Mean 0.35
Statistical Analysis 2: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to middle temporal gyrus activation (beta) on the semantic judgment fMRI task; Test type: Other — Null-hypothesis significance test; p = .412, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.24, 95% CI 2-sided [-0.34 to 0.81], Standard Error of Mean 0.29
Statistical Analysis 3: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to precuneus gyrus activation (beta) on the semantic judgment fMRI task; Test type: Other — Null-hypothesis significance test; p = .438, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = 0.31, 95% CI 2-sided [-0.48 to 1.09], Standard Error of Mean 0.40

12. Secondary Outcome: Relationship of Tau Burden to Resting-State Brain System Segregation
Description: Resting-state brain system segregation was computed on data collected from a separate resting-state scan using graph theory. System segregation is calculated as (Zw - Zb) / Zw, where Zw is the mean Fisher z-transformed r between nodes with the same system and Zb is the mean Fisher z-transformed r between nodes of one system to all nodes in other systems. Higher values indicate reduced node-node connectivity between systems relative to within-system connectivity. A score of 0 would reflect equal resting-state connectivity between nodes within the same functional system and between nodes of separate systems. Like all Z-scores, these scores typically range from -3 to 3. Higher scores are observed in younger adults than in older adults and may suggest a more youth-like brain, though higher scores are not objectively better. Systems were defined based on Power et al., (2011, Neuron) and more details on this measure are described in Chan et al. (2014, PNAS).
Time Frame: 1-year post study completion
Population: Participants with available data were analyzed. This sample excluded 2 statistical outliers.
Measure: Mean (Standard Deviation); unit: Z-score
Arm/Group | Follow up DLBS Participants
Number analyzed (Participants) | 105
Z-score | 0.58 (0.07)
Statistical Analysis 1: Comparison: Follow up DLBS Participants; Regression testing the relationship of temporal tau SUVR to resting-state system segregation; Test type: Other — Null-hypothesis significance test; p = .026, Regression, Linear — A priori threshold was two-sided 0.05. No adjustment for multiple comparisons; Adjusted for age, sex, and years of education; Slope = -1.13, 95% CI 2-sided [-2.12 to -0.14], Standard Error of Mean 0.50

ADVERSE EVENTS:
Time Frame: Day of visit (post-injection, pre-discharge) and follow-up call 48-72 hours post-injection
Description: The experimenter inquired about adverse events (AEs) during the time frames described above and, if AEs were reported, they filled out a log indicating the date/time, severity (mild, moderate, severe), possible relation to drug/procedure, action taken, and event resolution (e.g., resolved, ongoing).
Arm/Group | Follow up DLBS Participants
All-Cause Mortality (participants affected / at risk) | 0/125
Serious Adverse Events (participants affected / at risk) | 0/125
Other Adverse Events (participants affected / at risk) | 13/125
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Follow up DLBS Participants (N=125)
Elevated blood pressure (Blood and lymphatic system disorders) | 9 — AE resolved by 48-72 hour follow-up call.
Black dot in visual field (Eye disorders) | 1 — AE resolved by 48-72 hour follow-up call.
Muscle soreness in injection arm (Musculoskeletal and connective tissue disorders) | 1 — AE resolved by 48-72 hour follow-up call.
Neck rash (Skin and subcutaneous tissue disorders) | 1 — AE resolved by 48-72 hour follow-up call.
Diarrhea, drowsiness, nausea (General disorders) | 1 — AE resolved by 48-72 hour follow-up call.

LIMITATIONS AND CAVEATS:
Although several of these participants had an earlier PET-tau scan and we originally proposed to analyze longitudinal effects of tauopathy, a new PET scanner was implemented for this final wave of PET-tau data collection; preliminary analyses and discussions indicated the two scanners were not comparable and so we opted to focus on only this final wave of PET-tau data.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-18): https://cdn.clinicaltrials.gov/large-docs/44/NCT04080544/Prot_SAP_000.pdf
  • Informed Consent Form (2022-04-20): https://cdn.clinicaltrials.gov/large-docs/44/NCT04080544/ICF_001.pdf